CLINICAL TRIAL: NCT00542243
Title: A Phase III, Randomized, Double-Blind, Placebo Controlled Trial of PROSCAR in Men With Initial Negative Prostate Biopsies
Brief Title: A Trial of PROSCAR (Finasteride) Versus Placebo in Men With an Initial Negative Prostate Biopsy
Acronym: Prostress
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Merck Frosst Canada Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 07-0499-B; NCT00547079 (obsolete NCT alias)
Record Dates: First submitted 2007-10-09; First posted 2007-10-11 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-12

CONDITIONS: Enlarged Prostate
Keywords: enlarged prostate; finasteride
MeSH Terms: interventions — Finasteride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Finasteride (Active Comparator): The recommended dosage of PROSCAR© is one 5 mg tablet daily with or without food. If a tablet is missed at its usual time, an extra dose should not be taken. The next dose should be taken as usual.
  PROSCAR© 5 mg tablets are blue, apple-shaped; film coated with the code MSD 72 on one side and PROSCAR on the other. They will be provided in bottles of 35 tablets.
  Interventions: Drug: Finasteride
- Placebo (Placebo Comparator): Patient will receive a placebo comparator each day for 6 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Finasteride — Finasteride (5mg) will be given once per day for 6 months.
  Other Names: PROSCAR
  Arms: Finasteride
Drug: Placebo — Placebo will be given once a day for 6 months.
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess whether six months of daily finasteride (PROSCAR), following an initial negative prostate biopsy, will improve the detection of prostate cancer on repeat biopsy.

144 subjects with an initial negative prostate biopsy will be randomized to receive either finasteride or placebo for 6 months. The subjects will undergo a second prostate biopsy following drug intervention. PSA (prostate specific antigen) measurements, testosterone levels, and quality of life questionnaires will also be assessed during the study. The two groups will then be compared.

DETAILED DESCRIPTION:
5.0. Study Design and Treatment 5.1. Study Design This is a randomized, two-arm, double blind, placebo controlled study of daily PROSCAR® or placebo for 6 months in men with an initial negative prostate biopsy.

5.1.1. Biopsy The TRUS guided biopsy, to be carried out at Visit 4, will be performed by one physician. The biopsy will be performed as per the standard protocol at UHN, including 13-15 cores. The physician performing the biopsy will be blinded to the initial biopsy results and the PSA change over time. Before biopsy, a DRE will be performed. Aside from the standard biopsy scheme, suspicious areas on TRUS can be further biopsied. (e.g. a hypoechoic nodule).

5.2. Methods for Accrual and Randomization: Patients with an initial negative prostate biopsy that was performed at UHN and seen at the Prostate Center of the Princess Margaret Hospital will be considered for enrolment. Randomization by a random numbers table will be performed in blocks of 4 patients. After patients are deemed eligible for the study, the central office at Merck will be contacted and patient assignment given. The code will match the study drug label and the drug shipment will contain a blinded allocation envelope. The investigators, study participants and research coordinators will be blinded to the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Initial biopsy, performed at UHN, of at least 8 cores with no evidence of cancer (HGPIN or ASAP allowed)
* PSA < 20 ng/ml
* Able to swallow and retain oral medication
* Able to read and write (IPSS questionnaire is self-administered), understand instructions related to study procedures and to give written informed consent.

Exclusion Criteria:

* Glucocorticoids, except inhaled or topical, are not permitted within 3 months prior to visit one.
* Concurrent and previous use within the past 12 months of the following medications: Finasteride (PROSCAR, Propecia), Dutasteride (Avodart), Any other investigational 5 alpha-reductase inhibitors, Anabolic steroids, drugs with antiandrogenic properties.
* Participation in an investigational or marketed drug trial within the 30 days prior to the first dose of study drug or anytime during the study period.
* Abnormal liver function test (greater than 2 times the upper limit of normal) for alanine aminotransferase, aspartate aminotransferase, or alkaline phosphatase; or bilirubin > 1.5 times the upper limit of normal.
* Serum creatinine > 1.5 times the upper limit of normal.
* Any unstable serious co-existing medical conditions including but not limited to myocardial infarction, coronary bypass surgery, unstable angina, cardiac arrhythmias, clinically evident congestive heart failure, or cerebrovascular accident within 6 months prior to screening visit; uncontrolled diabetes or peptic ulcer disease which is uncontrolled by medical management.
* History of any illness (including psychiatric) that, in the opinion of the investigator, might confound the results of the study or pose additional risk to the subject.
* Known hypersensitivity to any 5 alpha-reductase inhibitor or to any drug chemically related to finasteride.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2008-02; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
The rate of prostate cancer at repeat TRUS (Transrectal Ultrasound) guided biopsy after 6 months of therapy with Finasteride/placebo. | 6 months

SECONDARY OUTCOMES:
Change in PSA parameters over time: a. PSA velocity b. PSA density c. Free/total PSA. | 6 months
TRUS at baseline and at the 6-month biopsy will be used to measure the total gland and transition zone volumes. | 6 months
TRUS nodule detection/visibility. | 6 months
Prostate vascularity as detected by Doppler ultrasound. | 6 months
Quality of life as tested by the IPSS (International Prostate Symptom Score). | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Finelli, MD MSc FRCSC, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Princess Margaret Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Kaplan SA, Ghafar MA, Volpe MA, Lam JS, Fromer D, Te AE. PSA response to finasteride challenge in men with a serum PSA greater than 4 ng/ml and previous negative prostate biopsy: preliminary study. Urology. 2002 Sep;60(3):464-8. doi: 10.1016/s0090-4295(02)01760-0. PMID 12350485
- [Background] Handel LN, Agarwal S, Schiff SF, Kelty PJ, Cohen SI. Can effect of finasteride on prostate-specific antigen be used to decrease repeat prostate biopsy? Urology. 2006 Dec;68(6):1220-3. doi: 10.1016/j.urology.2006.08.1070. Epub 2006 Dec 4. PMID 17141826
- [Background] Thompson IM, Chi C, Ankerst DP, Goodman PJ, Tangen CM, Lippman SM, Lucia MS, Parnes HL, Coltman CA Jr. Effect of finasteride on the sensitivity of PSA for detecting prostate cancer. J Natl Cancer Inst. 2006 Aug 16;98(16):1128-33. doi: 10.1093/jnci/djj307. PMID 16912265
- [Background] Thompson IM, Tangen CM, Goodman PJ, Lucia MS, Parnes HL, Lippman SM, Coltman CA Jr. Finasteride improves the sensitivity of digital rectal examination for prostate cancer detection. J Urol. 2007 May;177(5):1749-52. doi: 10.1016/j.juro.2007.01.071. PMID 17437804